CLINICAL TRIAL: NCT01186809
Title: Sequential Infusion of Unmanipulated Donor Lymphocytes and Cytokine Induced Killer (CIK)Cells After Allogeneic Stem Cell Transplantation
Brief Title: Cytokine Induced Killer (CIK) Cells In Leukemia Patients
Acronym: CIK2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Regional Hospital of Bolzano (Other); Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Rambaldi Alessandro, Prof, A.O. Ospedale Papa Giovanni XXIII
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eudract number: 2008-003185-26
Record Dates: First submitted 2010-08-10; First posted 2010-08-23 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Hematologic Malignancies
Keywords: hematologic malignancies (excluding Chronic Myeloid Leukemia)
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cytokine Induced Killer (Experimental): Sequential Infusion of Unmanipulated Donor Lymphocytes and Cytokine Induced Killer (CIK)
  Interventions: Biological: in vitro expanded Cytokine Induced Killer (CIK) cells

INTERVENTIONS:
Biological: in vitro expanded Cytokine Induced Killer (CIK) cells — Three infusions of donor Cytokine Induced Killer (CIK) cells will be administered according to a dose escalating program, starting 3 weeks after second Donor Lymphocyte Infusions (DLI). Cytokine Induced Killer administrations will be separated by 3 weeks intervals
  Other Names: patients will be offered Cytokine Induced Killer(CIK) cells.; Four combinations of escalating Cytokine Induced Killer (CIK) cells infusions will be provided, until the MTD will be defined.; Combination 1st CIK cells infusion 2nd CIK cells infusion 3rd CIK cells infusion; 1 1x106/Kg 1x106/Kg 5x106/kg; 2 1x106/Kg 5x106/kg 5x106/kg; 3 1x106/Kg 5x106/kg 10x106/kg; 4 5x106/kg 5x106/kg 10x106/kg

SUMMARY:
The purpose of the Phase IIA study are to:

1. define the safety profile
2. evaluate the efficacy of a sequential infusion of unmanipulated Donor Lymphocyte Infusions (DLI) and Cytokine Induced Killer (CIK) cells for the treatment of molecular, cytogenetic or hematologic relapse after hematopoietic stem cell transplantation and The progression free survival and the overall survival after the sequential infusion of Donor Lymphocyte Infusions (DLI) and Cytokine Induced Killer(CIK) cells.

DETAILED DESCRIPTION:
This study is an open-label, multicenter, exploratory phase IIA study to evaluate the safety (dose-finding) and efficacy of a sequential administration of donor derived unmanipulated DLI and in vitro expanded Cytokine Induced Killer(CIK) cells.

Two infusions of unmanipulated donor lymphocytes (1x106/Kg each) will be given with a minimum interval of 3 weeks. Three infusions of donor Cytokine Induced Killer (CIK) cells will be administered according to a dose escalating program, starting 3 weeks after second Donor Lymphocyte Infusions (DLI). In presence of grade 2 or more acute graft versus host disease(GVHD), the patient will not receive the next scheduled infusion. Only grade 4 acute graft versus host disease (aGVHD) is considered for the dose limiting toxicity (DLT). Once identified the maximally tolerated dose (MTD), this same combination of doses will be administered up to 24 patients in a two-stage minimax design.

Primary Endpoints

The primary endpoints of the Phase IIA study are:

1. the Maximally Tolerated Dose (MTD) - (safety end-point)
2. the cumulative incidence of molecular, karyotypic or haematologic responses at day +100 after the end of the cell therapy program - (efficacy end-point)

Secondary Endpoints Progression Free Survival (PFS) Progression Free Survival (PFS) will be defined as any evidence of molecular, cytogenetic or haematologic disease progression. Cytogenetic and/or molecular relapse will be defined where available as any evidence of a pre-transplant defined abnormality using conventional cytogenetics or FISH techniques or molecular probes. Assessments will be performed at 1 year after the end of the cell therapy program Overall Survival (OS) The Overall Survival(OS) will be assessed by 1 year after the end of the cell therapy program. For assessment of the Overall Survival (OS), events will be deaths for any causes, patients being censored if alive.

ELIGIBILITY:
Inclusion Criteria:

* Patients with haematologic malignancies (excluding chronic myeloid Leukemia- CML) with a molecular, cytogenetic or haematologic relapse after allogeneic transplantation.
* Patients with an available donor willing to donate peripheral blood lymphocytes
* Immunosuppression must be withdrawn at the beginning of the cell therapy program
* Written informed consent prior to any study procedures being performed

Exclusion Criteria:

* Donors positive for HIV, HBV or HCV, or unfit to undergo leukapheresis
* Patients with active acute or chronic Graft versus host disease (GvHD)
* Patients with rapidly progressive disease or not controlled by palliative supportive treatments including chemotherapy and with a life expectancy less than 8 weeks
* Patients with severe psychiatric illness or any disorder that compromises ability to give truly informed consent for participation in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-07; Primary Completion 2016-09 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro AR Rambaldi, Professor, Principal Investigator — Azienda Ospedaliera Papa Giovanni XXIII (Former:Ospedali Riuniti di Bergamo)
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Papa Giovanni XXIII (Former:Ospedali Riuniti di Bergamo) Bergamo, Bergamo
  - Ospedale Centrale di Bolzano, Bolzano
  - Ospedale San Gerardo, Monza

IPD SHARING:
Plan to Share IPD: Yes
final report

REFERENCES:
- [Result] Introna M, Franceschetti M, Ciocca A, Borleri G, Conti E, Golay J, Rambaldi A. Rapid and massive expansion of cord blood-derived cytokine-induced killer cells: an innovative proposal for the treatment of leukemia relapse after cord blood transplantation. Bone Marrow Transplant. 2006 Nov;38(9):621-7. doi: 10.1038/sj.bmt.1705503. Epub 2006 Sep 18. PMID 16980990
- [Result] Introna M, Borleri G, Conti E, Franceschetti M, Barbui AM, Broady R, Dander E, Gaipa G, D'Amico G, Biagi E, Parma M, Pogliani EM, Spinelli O, Baronciani D, Grassi A, Golay J, Barbui T, Biondi A, Rambaldi A. Repeated infusions of donor-derived cytokine-induced killer cells in patients relapsing after allogeneic stem cell transplantation: a phase I study. Haematologica. 2007 Jul;92(7):952-9. doi: 10.3324/haematol.11132. PMID 17606446
- [Result] Capelli C, Salvade A, Pedrini O, Barbui V, Gotti E, Borleri G, Cabiati B, Belotti D, Perseghin P, Bellavita P, Biondi A, Biagi E, Rambaldi A, Golay J, Introna M. The washouts of discarded bone marrow collection bags and filters are a very abundant source of hMSCs. Cytotherapy. 2009;11(4):403-13. doi: 10.1080/14653240902960437. PMID 19462317
- [Result] Introna M, Pievani A, Borleri G, Capelli C, Algarotti A, Mico C, Grassi A, Oldani E, Golay J, Rambaldi A. Feasibility and safety of adoptive immunotherapy with CIK cells after cord blood transplantation. Biol Blood Marrow Transplant. 2010 Nov;16(11):1603-7. doi: 10.1016/j.bbmt.2010.05.015. Epub 2010 Jun 1. PMID 20685246

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 74 patients were enrolled in the study from July 2009 to September 2016
Groups:
- Cytokine Induced Killer: Sequential Infusion of Unmanipulated Donor Lymphocytes and Cytokine Induced Killer (CIK)
  in vitro expanded Cytokine Induced Killer (CIK) cells: Three infusions of donor Cytokine Induced Killer (CIK) cells will be administered according to a dose escalating program, starting 3 weeks after second Donor Lymphocyte Infusions (DLI). Cytokine Induced Killer administrations will be separated by 3 weeks intervals
  This is a phase IIA study to evaluate the safety (dose-finding) and efficacy of a sequential administration of donor derived unmanipulated DLI and in vitro expanded CIK cells. Two infusions of unmanipulated donor lymphocytes (1x106/Kg each) will be given with a minimum interval of 3 weeks. Three infusions of donor CIK cells will be administered according to a dose escalating program, starting 3 weeks after second DLI. CIK administrations will be separated by 3 weeks intervals. Standard treatment with unmanipulated DLI will be offered to patients refusing the proposal.
Period: Overall Study
Arm/Group | Cytokine Induced Killer
Started | 73
Completed | 43
Not Completed | 30
Not completed — Death | 30

BASELINE CHARACTERISTICS:
Arm/Group | Cytokine Induced Killer
Number analyzed (Participants) | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 58
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 39
Region of Enrollment [Number; unit: participants]
  Italy | 73

OUTCOME MEASURES:

1. Primary Outcome: Safety Measures
Description: The occurrence of a grade 4 acute graft versus host disease (GVHD), judged to be related to the study medication. Grading and staging will be performed using the Glucksberg scale
Time Frame: Clinical response was measured at 100 days after the completion of the cell therapy program.
Measure: Number; unit: participants
Arm/Group | Cytokine Induced Killer
Number analyzed (Participants) | 73
participants | 0

2. Secondary Outcome: Efficacy Measures
Description: The proportion of patients achieving a complete, a partial or a hematologic improvement in responses to the experimental infusion of cytokine induced killer (CIK)cells
Time Frame: The clinical response will be registered at day +100 after the last Cytokine Induced Killer (CIK) cell infusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: three years;
Arm/Group | Cytokine Induced Killer
All-Cause Mortality (participants affected / at risk) | 31/73
Serious Adverse Events (participants affected / at risk) | 8/73
Other Adverse Events (participants affected / at risk) | 16/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytokine Induced Killer (N=73)
aGVHD grade III; IV (Gastrointestinal disorders) | 5 (5) — acute graft versus host disease
hemolitic anemia (Blood and lymphatic system disorders) | 1 (1) — severe hemolitic anemia
severe chronic GVHD (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytokine Induced Killer (N=73)
aGvHD (Skin and subcutaneous tissue disorders) | 7 (7) — grade 1-2 acute graft versus host disease
cGvHD (Skin and subcutaneous tissue disorders) | 9 (9) — mild and moderate chronic graft versus host disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes